CLINICAL TRIAL: NCT03526133
Title: Validation of a Wireless Wearable Sensor Using Mobile Technology and Cloud Computing for the Diagnosis of Sleep Apnea
Brief Title: Validation of Sleep Apnea Diagnosis Device
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Biologix Sistemas Ltda (Unknown)
Responsible Party: Sponsor
Other Study IDs: 70485317.0.0000.0068
Record Dates: First submitted 2018-04-12; First posted 2018-05-16 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2018-07

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; polygraph; home sleep apnea test (HSAT); apnea hypopnea index (AHI); oxygen desaturation index (ODI); portable monitor; sleep actimetry; snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) and wireless sensor Oxistar — Monitoring the apnea-hypopnea index (AHI) derived from PSG and the oxygen desaturation index (ODI) obtained by the Oxistar.

SUMMARY:
Obstructive sleep apnea (OSA) is common and largely underdiagnosed disease. The standard method for the diagnosis of OSA is a complete night polysomnography (PSG). Simple methods for OSA diagnosis are necessary. The overnight oximetry with the oxygen desaturation index (ODI) has been largely investigated as a diagnostic test for OSA but its accuracy remains undefined. The aim of our study is to evaluate if an wireless polygraph (Oxistar) is accurate to diagnosis OSA in patients referred to a Sleep Lab.

DETAILED DESCRIPTION:
Consecutive patients referred to the sleep laboratory with suspected diagnosis of OSA underwent in-laboratory polysomnography (PSG) and simultaneously wireless polygraph. The PSG oximeter and the wireless polygraph were worn on different fingers of the same hand. All sleep studies were reviewed by one blind investigator according the 2017 American Academy of Sleep Medicine recommendations. The number of desaturations from wireless polygraph at the 3 predefined threshold levels (of ODI-2%, ODI-3%, or ODI-4%) was derived automatically using proprietary algorithm. Moderate to severe OSA was defined as AHI ≥ 15 events/h. The diagnostic accuracy of ODI-2%, 3%, and 4% for the diagnosis of moderate-severe OSA were calculated for cut-off values from 1 to 20 desaturation events/h. The sleep actimetry was compared with the sleep stages from PSG, most of the statistical metrics applied for diagnosis were used to evaluate the applicability of this proposed method. Finally, the snoring events computed by the smartphone application were compared with the events heard by a specialist and the statistical comparison metrics were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* referred by medical staff for an overnight assessment for suspected sleep apnea

Exclusion Criteria:

* polysomnography for the CPAP titration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to a university-based tertiary sleep referral centre.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Night during the polysomnography exam
  Sensitivity of Oxistar device to detect apnea events compared to gold-standard polysomnography
Specificity | Night during the polysomnography exam
  Specificity of Oxistar device to detect apnea events compared to gold-standard polysomnography
Area under the curve (AUC) | Night during the polysomnography exam
  AUC from ROC curves reflects the accuracy of Oxistar device to detect apnea events compared to gold-standard polysomnography
Bland-Altman Graph | Night during the polysomnography exam
  The Bland-Altman graph evaluates the "agreement" between the gold-standard polysomnography and Oxistar device
Interclass Correlation Coefficient (ICC) | Night during the polysomnography exam
  ICC measures the reliability of measurements or ratings between the gold-standard polysomnography and Oxistar device

SECONDARY OUTCOMES:
Sleep Actigraphy | Night during the polysomnography exam
  Actigraphy is the continuous measurement of activity or movement with the use of a small device called an actigraph. Periods of movement suggest wakefulness while those of relative stillness would likely correspond to sleep or quiescence. The Oxistar has a embeded actigraph whose data will be compared with the sleep stage scoring from polysomnography (PSG), the gold standard for sleep assessment. Epoch-by-epoch (30 seconds) agreement between the actigraph and PSG will be assessed by calculating sensitivity, specificity, accuracy, area under the curve (AUC), Bland-Altman graph and interclass correlation coefficient (ICC)
Number of snoring events per hour of register (snoring/h) | Night during the polysomnography exam
  Snoring is one of the signs suggestive of obstructive sleep apnea and has recently been considered as having great diagnostic potential. The smartphone application (app) through microphone performs the recording and the characteristics extraction of the patient's audio during sleep (register time). A multilayer perceptron (MPL) neural network classifies the event as snoring or non-snoring. Lastly, the amount of snoring occured is accounted and divided by the register time leading to the number of snoring/h. The agreement between snoring/h measured by the app and the heard by a specialist will be assessed by calculating sensitivity, specificity, accuracy and area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi-Filho, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Incor - Heart Institute, Sleep Laboratory, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinheiro GDL, Cruz AF, Domingues DM, Genta PR, Drager LF, Strollo PJ, Lorenzi-Filho G. Validation of an Overnight Wireless High-Resolution Oximeter plus Cloud-Based Algorithm for the Diagnosis of Obstructive Sleep Apnea. Clinics (Sao Paulo). 2020 Nov 27;75:e2414. doi: 10.6061/clinics/2020/e2414. eCollection 2020. PMID 33263626